CLINICAL TRIAL: NCT03395366
Title: Improving Outcomes for Hemodialysis Patients by Addressing Poor Health Related Quality of Life With Cognitive Behavioral Strategies
Brief Title: Improving Outcomes for Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Satellite Healthcare (Other)
Responsible Party: Principal Investigator, Shayan Shirazian, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AAAR6257
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Quality of Life; End Stage Renal Disease
Keywords: Hemodialysis; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: The study will be designed as a 16-week randomized controlled trial in which 40 subjects on hemodialysis with below average HrQOL will be assigned to one of two educational interventions.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Multifaceted Educational / Cognitive Behavioral Intervention
  Interventions: Other: Multifaceted Educational / Cognitive Behavioral Intervention
- Group 2 (No Intervention): Standard of Care + Dialysis Education without the Cognitive Behavioral component

INTERVENTIONS:
Other: Multifaceted Educational / Cognitive Behavioral Intervention — The intervention includes 8 to 12 one-on-one sessions over a 12-week period, run by a licensed social worker (LSW) with experience delivering therapy. Curriculum will introduce education relevant for self-management and consists of prepared slides, handouts & worksheets. The education was designed based on slides developed and published online by the national kidney foundation and the national kidney disease education program. The curriculum was designed to be understandable by all potential subjects, including those with low literacy levels. Sessions will incorporate behavior-based activities designed to deliver education about and improve upon medication adherence, diet, exercise, and coping. These activities, based around CB strategies such as cognitive restructuring and behavior shaping, will include review of self-management logs, goal setting, creation of treatment plan, problem-solving techniques, reinforcing techniques, and coping with ESRD.
  Arms: Group 1

SUMMARY:
End stage renal disease (ESRD) affects approximately 700,000 Americans of which approximately 400,000 are on life-saving hemodialysis therapy. Hemodialysis can take a physical and emotional toll on patients, and most patients on hemodialysis describe poor quality of life. Patients on hemodialysis have worse health related quality of life (HrQOL) than patients with any other chronic illness including cancer and congestive heart failure. This poor quality of life can affect how well these patients manage their own health or their self-care, and can ultimately lead to poor health outcomes. Despite this, there are no commonly used programs to improve quality of life or self-care for patients on hemodialysis. The investigators have developed a simple 3-step program to improve quality of life and self-care for patients on hemodialysis. The first step involves presenting quality of life scores to the dialysis health care team so that a program can be designed. The second step involves 8-12 education sessions combined with behavioral training designed to improve quality of life and self-care. The final step is monthly re-evaluation of progress. In this study, the investigators will test this 3-step program, compared to dialysis education alone, to see if it improves quality of life and self-care. By improving quality of life and self-care the investigators believe patient outcomes including hospitalizations will improve.

DETAILED DESCRIPTION:
Hemodialysis (HD) patients have worse health related quality of life (HrQOL) than patients with any other chronic illness. In this population, poor quality of life and depressive symptoms (a major component of HrQOL) are associated with medication non-compliance, dietary indiscretion, interdialytic weight gain, and missed dialysis. These associations likely explain the link between low HrQOL scores and adverse medical outcomes. Even small decrements in HrQOL score are associated with an increased risk of hospitalizations and mortality. Moreover, depressive symptoms occur in one-third of HD patients and are themselves associated with increased hospitalizations and with a 1.5 times higher mortality risk.

To address poor HrQOL in HD patients, the Centers for Medicare Services (CMS) mandated its screening on a regular basis in all HD patients. However, CMS has not mandated how to present HrQOL results to key HD providers, or how to treat those with poor HrQOL. Nor are there widely applied methods of doing so. Although prior interventions in HD patients have improved quality of life and self-management, these interventions were limited by poor patient and physician adoption, a lack of reproducible methods, selective inclusion and exclusion criteria and a lack of translatability. To date there are no widely adopted interventions to improve quality of life in this population. Thus, it is not surprising that, HrQOL scores remain unchanged in 8 years since the CMS mandate. In sum, HrQOL survey results have not been applied in a manner that makes a difference for patients.

Cognitive behavioral therapy (CBT) is a structured psychotherapy intervention designed to address and treat dysfunctional cognitions, negative emotions and maladaptive behaviors. In patients with chronic illness, CBT has been adapted to successfully improve adherence to self-management behaviors. In patients with ESRD, several studies have used cognitive behavioral strategies to improve self-management, quality of life, and depressive symptoms. These studies however were limited by high drop-out rates and a lack of translatability. To date, cognitive behavioral (CB) strategies are not routinely used in the care of ESRD patients.

The investigators have developed a simple, translatable 3-step intervention to improve poor HrQOL in hemodialysis patients. The first step is a one-page dashboard that presents actionable HrQOL data to key stakeholders (social workers, nutritionists, primary nurses, nurse-practioners, physicians, patients and family members) during monthly case conference. The second step is a treatment approach that combines self-management education with CB strategies through 8-12 simple sessions delivered chair-side over 12 weeks. These sessions are designed to be delivered by unit social workers and are highly translatable to other US hemodialysis units. The final step is monthly re-evaluation at clinical case conference where patient progress will be assessed and the dashboard and behavioral-education sessions refined. Each step of the intervention was designed to be highly translatable to current hemodialysis care. The dashboard utilizes data that is currently checked, the treatment sessions are delivered by social workers that are already employed at hemodialysis centers and re-evaluation occurs during monthly case conference sessions that are already being held.

The investigators hypothesize that implementing their multi-faceted intervention will improve HrQOL, depressive symptoms and self-management, and will be immediately translatable to other US hemodialysis units. Therefore, the investigators propose to conduct a 16-week randomized controlled trial in 40 subjects on hemodialysis with poor HrQOL to test the impact of the intervention on these outcomes. The primary outcome, Kidney Disease Quality of Life Short Form 36 (KDQOL-36™) survey scores, will be measured at 0, 8, and 16 weeks. Through end-of-study focus groups, the investigators will refine the intervention and help translate our intervention into practice. Additionally, the investigators will develop a translatable toolbox that will give step-by-step instructions on how to implement our intervention at other US hemodialysis units. Finally, the investigators will explore the effect of our intervention on hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients on hemodialysis for at least 3 months
* Most recent 36-question Kidney Disease Quality of Life (KDQOL-36), Physical Component Summary (PCS), or Mental Component Summary (MCS) score below 50
* KDQOL-36 burden of disease score 80
* Expected survival 6 months
* English-speaking

Exclusion Criteria:

* Bipolar or Psychotic disorder
* Moderate or severe cognitive impairment as determined by the hemodialysis staff or documented in the electronic medical record (EMR)
* Severe vision or hearing impairment
* Drug or alcohol dependence
* Active suicidal ideation or a history of suicide attempt (determined based on screening patient health questionnaire-9 and EMR)
* Current participation in a behavioral or education treatment program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Change in score on Kidney Disease Quality of Life Short Form 36 (KDQOL-36™) | 0 weeks, 8 weeks, 16 weeks
  The investigators will summarize the average changes from pre to post for each treatment arm via means (±SD) and 95% confidence intervals and estimate the effect of our intervention by estimating a linear model for each post-treatment score, adjusting for pre-treatment score and treatment arm (i.e. an ANCOVA model).

CONTACTS AND LOCATIONS:
Overall Officials: Shayan Shirazian, MD, Principal Investigator — Columbia University
Locations (1):
- DaVita Columbia University Dialysis, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shirazian S, Smaldone AM, Jacobson AM, Fazzari MJ, Weinger K. Improving quality of life and self-care for patients on hemodialysis using cognitive behavioral strategies: A randomized controlled pilot trial. PLoS One. 2023 May 4;18(5):e0285156. doi: 10.1371/journal.pone.0285156. eCollection 2023. PMID 37141225